CLINICAL TRIAL: NCT06874049
Title: Oral Versus Vaginal Misoprostol Solution Among Pregnant Women Undergoing Induction of Labor At Ain Shams University Maternity Hospital a Randomized Controlled Trial
Brief Title: Comparison Between Vaginal Misoprostol Gel and Oral Misoprostol Solution in Induction of Labor
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Hagar Muhammad Abdulfattah Muhammad (Other)
Responsible Party: Sponsor-Investigator, Hagar Muhammad Abdulfattah Muhammad, Obstetrics and Gynecology resident, Ain Shams Maternity Hospital
Organization: Ain Shams Maternity Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1525
Record Dates: First submitted 2025-03-05; First posted 2025-03-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Cervical Ripening and Induction of Labor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- vaginal misoprostol solution (Experimental): the vaginal solution will be prepared by complete crushing of one misoprostol 200 µg tablet into powder then adding the powder into a clean urine specimen cup then adding 20 cc of KY gel measured by a 20 ml syringe then mix the contents together to ensure adequate distribution of the powder , each patient will receive only 2.5cc of the mixture vaginally (inserted into the posterior fornix,) by using medical 3ml syringes equal to 25 mcg misoprostol 4 hourly according to International Federation of Gynecology and Obstetrics (FIGO2023) and remain recumbent for 10-20 minutes.
  Interventions: Drug: Vaginal misoprostol
- oral misoprostol solution (Active Comparator): the first group the solution will be prepared by dissolving one 200 µg tablet in 200 ml of tap water , each member will receive 25 cc misoprostol solution equal to 25 mcg misoprostol 2 hourly according to International Federation of Gynecology and Obstetrics (FIGO2023).
  Interventions: Drug: Oral misoprostol solution (OMS)

INTERVENTIONS:
Drug: Vaginal misoprostol — the vaginal misoprostol solution will be prepared by complete crushing of one misoprostol 200 µg tablet into powder then adding the powder into a clean urine specimen cup then adding 20 cc of KY gel measured by a 20 ml syringe then mix the contents together to ensure adequate distribution of the powder , each patient will receive only 2.5cc of the mixture vaginally (inserted into the posterior fornix,) by using medical 3ml syringes equal to 25 mcg misoprostol 4 hourly according to International Federation of Gynecology and Obstetrics (FIGO2023) and remain recumbent for 10-20 minutes
  Arms: vaginal misoprostol solution
Drug: Oral misoprostol solution (OMS) — the solution will be prepared by dissolving one 200 µg tablet in 200 ml of tap water , each member will receive 25 cc misoprostol solution equal to 25 mcg misoprostol 2 hourly according to International Federation of Gynecology and Obstetrics (FIGO2023)
  Arms: oral misoprostol solution

SUMMARY:
The goal of this clinical trial is to study the efficacy of vaginal versus oral misoprostol solution in cervical ripening for induction of labor.

The main questions it aims to answer is : is Vaginal misoprostol solution as effective as oral misoprostol solution for induction of labor? Researchers will compare oral Misoprostol Solution and vaginal misoprostol solution prepared by KY gel Participants will then be randomized into two groups using a computer-generated randomization list , the first group will receive oral solution equal to 25 microgram misoprostol every 2 hours while the second group will receive 25 microgram vaginal misoprostol solution every 4 hours The cervix will be assessed and scored at each examination. They will be reviewed before the stipulated time if they were contracting. The administration of the drugs will be discontinued when a favorable cervix is diagnosed (modified Bishop score ≥6 ) or 24 hours of study drug had been given.

ELIGIBILITY:
Inclusion Criteria:

1. Women with a singleton pregnancy.
2. Cephalic presentation.
3. Age range: 18-40 years.
4. Gestational age between 36 and 42 weeks.
5. Intact fetal membranes.
6. Absence of spontaneous uterine contractions.
7. Non favorable cervix (Bishop score ≤ 5).
8. A reactive non stress test in case of positive fetal life.

Exclusion Criteria:

1. History of cesarean section or uterine scars
2. Grand Multipara P ≥5
3. Known fetal non-cephalic presentation
4. Any known allergy to misoprostol.
5. Multiple pregnancy
6. Contraindication to vaginal delivery.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-02-26 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
The primary outcome measure is induction to cervical ripening (Bishop score ≥6) time interval. | 24 hours max

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams university Maternity Hospital, Cairo, Egypt